CLINICAL TRIAL: NCT07055828
Title: Nebulized Versus Intravenous Ketamine as Prophylaxis Against Spinal Anesthesia-induced Shivering and Hemodynamic Changes: A Placebo-controlled Prospective Study
Brief Title: Nebulized vs. IV Ketamine in Preventing Shivering Post Spinal Anesthesia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Lotfy, Assistant Professor of Anesthesia, Pain Management and Surgical ICU, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 36264PR1219/5/25
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Post Spinal Anesthesia Shivering
MeSH Terms: interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group P (Placebo) (Active Comparator): Patients in this group met the study's inclusion criteria and received inactive solutions (saline) both through nebulization and intravenously, serving as a control.
  Interventions: Drug: Normal Saline; Drug: Saline Inhalants
- Group NK (Nebulized Ketamine) (Active Comparator): Patients in this group met the study's inclusion criteria and received ketamine via a nebulizer at a specific dose. They also received intravenous saline as a placebo.
  Interventions: Drug: Intranasal ketamine; Drug: Normal Saline
- Group IVK (Intravenous Ketamine) (Placebo Comparator): Patients in this group met the study's inclusion criteria and received ketamine intravenously as a prophylactic drug before spinal anesthesia. They also received nebulized saline as a placebo.
  Interventions: Drug: Ketamine; Drug: Saline Inhalants

INTERVENTIONS:
Drug: Ketamine — Patients received IV ketamine 0.25 mg/kg before Spinal anesthesia as a prophylactic drug
  Arms: Group IVK (Intravenous Ketamine)
Drug: Intranasal ketamine — Patients received nebulized ketamine at a dose of 0.75 mg/kg adjusted to 5 ml by adding normal saline to be inhaled through a breath-actuated nebulizer
  Arms: Group NK (Nebulized Ketamine)
Drug: Normal Saline — Patients received Intravenous Normal saline
  Arms: Group NK (Nebulized Ketamine); Group P (Placebo)
Drug: Saline Inhalants — Patients received nebulized Saline
  Arms: Group IVK (Intravenous Ketamine); Group P (Placebo)

SUMMARY:
Shivering is an involuntary muscle activity, often triggered by hypothermia, that can occur after anesthesia. This is known as postanesthetic shivering (PAS) and is a common issue that increases oxygen demand, raises the risk of low oxygen levels, and can lead to complications after surgery.

Spinal anesthesia (SA) is a popular choice due to its quick action and effective numbing. However, it's frequently linked to shivering during and after the procedure.

To combat PAS, various methods have been used. Non-pharmacological approaches like insulation, continuous warming, and temperature management have been shown to reduce low body temperature during surgery and decrease shivering and complications afterward, aiding recovery.

Pharmacologically, certain medications can help. Intrathecal meperidine or intravenous (IV) ketamine are effective in preventing PAS. Intrathecal midazolam can also reduce shivering, unlike fentanyl. Additionally, IV ketamine infusion can lower the incidence of low blood pressure and shivering in patients receiving SA. Low-dose ketamine combined with dexmedetomidine, or dexmedetomidine alone, have also shown similar effectiveness in reducing shivering and postoperative nausea and vomiting during SA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were assigned for Inguinal Hernia hernioplasty;
* Patients free of exclusion criteria were enrolled in the study.

Exclusion Criteria:

* Patients who were on the American Society of Anesthesiologists Physical Status classification (ASA) grade >II;
* Patients with body mass index (BMI) >30 kg/m²;
* Patients with Upper respiratory tract diseases;
* Patients with spinal deformities or diseases;
* Patients with coagulopathy, or allergies to the drugs used;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Nebulized Ketamine on Post-Anesthesia Shivering (PAS) Incidence and Severity | 56 days
  This Study asses the effectiveness of the administered therapy in controlling Post-Anesthesia Shivering (PAS) as a reduction in both its incidence and severity. Specifically, effective control is indicated by a Bedside Shivering Assessment Score (BSAS) of less than 2 within the initial 60 minutes post-therapy, alongside a reduction in other associated adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El Gharbyia, Egypt